CLINICAL TRIAL: NCT04877652
Title: DR REGISTRY: Prospective Observational Study of Decongestion in Acute Heart Failure Patients With Insufficient Response to Diuretics
Brief Title: DR REGISTRY: Prospective Observational Study of ADHF Patients With Insufficient Response to Diuretics
Status: Completed | Type: Observational
Sponsor: Revamp Medical Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIS-D-02
Record Dates: First submitted 2021-04-19; First posted 2021-05-07 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Acute Decompensated Heart Failure
Keywords: ADHF
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ADHF patients: Patients with acute decompensated heart failure (ADHF) having insufficient response to diuretic therapy following a dose escalation protocol in keeping with AHA guidelines for the management of heart failure.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Standard of care — Standard medical treatment of ADHF patients deemed to have insufficient diuretic response.

SUMMARY:
The study objective is to observe and measure clinical outcomes, urine output, and safety events occurring during standard medical treatment of ADHF patients deemed to have insufficient diuretic response.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is >18 and < 85 years of age.
2. Subject is hospitalized with primary diagnosis of ADHF.
3. N-terminal-pro-brain natriuretic peptide (NT-proBNP) ≥1,600 pg/m or BNP≥400 pg/mL.
4. Evidence of fluid overload as indicated by 2 or more of the following criteria:

   1. peripheral edema ≥ 2+
   2. radiographic pulmonary edema or pleural effusion
   3. enlarged liver or ascites
   4. pulmonary rales or paroxysmal nocturnal dyspnea, or orthopnea
   5. Jugular venous distention > 7 cmH2O
5. Subject insufficiently responds to IV diuretic therapy

Exclusion Criteria:

1. Systolic blood pressure <90 mmHg at the time of screening.
2. Acute myocardial infarction or acute coronary syndrome or cardiogenic shock or pleural synthesis within past 7 days or cardiovascular intervention within past 4 days.
3. Known LVEF < 15% by echocardiography within 1 year prior to enrolment.
4. Complex congenital heart disease (e.g., Tetralogy of Fallot subjects, single ventricle physiology).
5. Known active myocarditis, hypertrophic obstructive cardiomyopathy, constrictive pericarditis or cardiac tamponade.
6. Severe Aortic valvular disorder (i.e., hemodynamically relevant valvular diseases such as severe stenosis \severe regurgitation) or Severe mitral disease with planned intervention.
7. Evidence of active systemic infection documented by either one of the following: fever >38°C/100°F, or ongoing uncontrolled infection (i.e., inflammatory parameters not decreasing despite > 48 hours of antibiotic treatment).
8. Moribund subject or subject with severe or deteriorating damage in more than 3 critical body systems, based on investigator's clinical judgement.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Heart Failure Patients with Insufficient Response to Diuretics
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Events | 30 days
  SAEs (including MACE) post enrollment based on CEC adjudication.
Serum Creatinine | Baseline [T=0] and 48 hours
  Change in level
Urine Output | Baseline [T=0-12h] and through 24 hours [T=12-36h]
  Change in the rate

OTHER OUTCOMES:
Dyspnea | Baseline [T=0] and 48 hours
  Change in dyspnea score using the Likert scale (score ranges from -3 to +3, higher score means better improvement)
Peripheral Edema | Baseline [T=0] and 48 hours
  Change in score (ranges from none/0 to +4)
Length of hospitalization | through follow-up period completion (up to 60 days)
  Length of current hospitalization (resolution of acute heart failure condition)
Heart Failure Readmission | Baseline through 30 days
  Time to readmission due to HF, up to 30 days

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Weill Cornell, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Montefiore Medical Center - Moses Campus, New York, New York
  - St Francis Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided